CLINICAL TRIAL: NCT05162742
Title: Does Colchicine Reduce Progression of Aortic Valve Stenosis?
Brief Title: Colchicine and Inflammation in Aortic Stenosis
Acronym: CHIANTI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112719
Record Dates: First submitted 2021-11-16; First posted 2021-12-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Calcification; Inflammation; Calcification; Cardiovascular Diseases
Keywords: Aortic Stenosis; Inflammation
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve, Calcification of; Inflammation; Calcinosis; Cardiovascular Diseases | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): 75 patients will receive colchicine tablets
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): 75 patients will receive placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — ATC: M04AC01
  Arms: Colchicine
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
Aortic stenosis (AS) is the most common valvular heart disease in the developed world. Once symptomatic, untreated patients have a poor prognosis with five-year survival rate of 25%. Once at an advanced stage, AS will lead to the development of left ventricle hypertrophy, and eventually heart failure and death. At-present, there is no effective medical therapy for aortic stenosis. Current management of patients with AS consists of 'watchful waiting'. Valve replacement is needed when these patients (often acutely) become symptomatic. Recent studies have shown that inflammatory processes with similarities to atherosclerosis play an important role in AS. Therefore, we hypothesize that treatment with anti-inflammatory therapy, in the form of colchicine, could reduce the progression of AS. If positive, this trial will be the first to provide a potential therapeutic option for millions of people world-wide with AS.

ELIGIBILITY:
Inclusion Criterion:

• Asymptomatic moderate aortic valve stenosis on recent (<6 months) echocardiography (based on peak velocity, mean gradient, aortic valve area). The severity of AS will be quantified according to current EACVI / ASE guidelines.

Exclusion Criteria:

* Heavily calcified aortic valve on echocardiography (defined as grade 4 calcification: extensive thickening/calcification of all cusps as described in the articles by Rosenhek et al.);
* a planned aortic valve replacement in the next six months;
* severe mitral valve stenosis (MVA < 1cm2);
* severe mitral or aortic valve regurgitation;
* rheumatic aortic valve disease;
* bicuspid aortic valve;
* valvular disease due to history of chest radiation;
* left ventricular dysfunction (LVEF < 35%);
* renal impairment (eGFR <30 ml/min/1.73m2);
* patients aged <50 and >80 years;
* pre-existing chronic gastro-intestinal complaints which may obscure signs of colchicine intolerance;
* child-bearing potential without the use of contraception;
* use of CYP3A4 (e.g. verapamil) or P-glycoprotein inhibitors;
* use of bisphosphonate or denosumab;
* chronic use of immunosuppressants or anti-inflammatory drugs including colchicine and NSAID's (excl. acetylsalicylic acid);
* active or chronic liver disease;
* the presence of a pacemaker or internal cardiac defibrillator;
* life expectancy <2 years.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in aortic valve calcium score | Baseline and 24 months
  Change in aortic valve calcium score measured by computed tomography aortic valve calcification (CT-AVC).

SECONDARY OUTCOMES:
Aortic valve 18F-NaF uptake | Baseline and 24 months
  Difference in aortic valve 18F-NaF uptake of the aortic valve using positron emission tomography (PET) between baseline and end of study.
Change in echocardiographic parameter for aortic stenosis | Baseline, 12 months and 24 months
  Determined by change in peak velocity (m/s)
Adverse Outcomes | Baseline and 24 months
  Determine the effect of colchicine on calcified aortic stenosis related adverse outcomes (cardiac death, myocardial infarction, stroke, (hospitalization for) heart failure and aortic valve replacement).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, The Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammadnia N, Vestjens LTW, Craig NJ, Tijssen JGP, Knol RJJ, Lazarenko SV, Duffels MGJ, Jaspers Focks J, Hemels MEW, Oving I, Schalkx HJ, Eikelboom JW, Cetinyurek-Yavuz A, Aarntzen EHJG, Dey D, Slomka PJ, Nijveldt R, Riksen NP, van Royen N, Honigberg MC, Dweck MR, Cornel JH, El Messaoudi S. The effects of low-dose colchicine on the progression of aortic valve stenosis: Rationale, design, and baseline characteristics of the Colchicine and Inflammation in Aortic Stenosis (CHIANTI) trial. Am Heart J. 2025 Dec;290:297-309. doi: 10.1016/j.ahj.2025.07.010. Epub 2025 Jul 12. PMID 40659197